CLINICAL TRIAL: NCT05158998
Title: Impact of Propofol Versus Sevoflurane on Incidence of Postoperative Delirium in Elderly Patients After Spine Surgery: a Randomized Controlled Trial
Brief Title: Impact of Propofol Versus Sevoflurane on Incidence of Postoperative Delirium in Elderly Patients After Spine Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: QianfoshanH PSPOD
Record Dates: First submitted 2021-11-18; First posted 2021-12-15 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Delirium in Old Age; Anaesthetic
Keywords: delirium; spine surgery; anaesthetic; propofol; sevoflurane
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Other): For patients in the propofol group, anaesthesia will be maintained with propofol infusion(target controlled infusion), of which the target concentration will be adjusted to maintain the BIS value between 40 and 60. Analgesia will be maintained with remifentanil(0.1-0.5ug/(kg.min)), muscle relaxation will be maintained with atracurium(10ug/(kg.min)). Propofol infusion will be stopped at the end of surgery.
  Interventions: Drug: propofol infusion
- sevoflurane group (Other): For patients in the sevoflurane group, anaesthesia will be maintained with sevoflurane inhalation, of which the concentration will be adjusted to maintain the BIS value between 40 and 60. Analgesia will be maintained with remifentanil(0.1-0.5ug/(kg.min)), muscle relaxation will be maintained with atracurium(10ug/(kg.min)). Sevoflurane inhalation will be stopped at the end of surgery.
  Interventions: Drug: sevoflurane inhalation

INTERVENTIONS:
Drug: propofol infusion — For patients in the propofol group, anaesthesia will be maintained with propofol infusion(target controlled infusion), of which the target concentration will be adjusted to maintain the BIS value between 40 and 60. Analgesia will be maintained with remifentanil(0.1-0.5ug/(kg.min)), muscle relaxation will be maintained with atracurium(10ug/(kg.min)).Propofol infusion will be stopped at the end of surgery.
  Arms: propofol group
Drug: sevoflurane inhalation — For patients in the sevoflurane group, anaesthesia will be maintained with sevoflurane inhalation, of which the concentration will be adjusted to maintain the BIS value between 40 and 60. Analgesia will be maintained with remifentanil(0.1-0.5ug/(kg.min)), muscle relaxation will be maintained with atracurium(10ug/(kg.min)). Sevoflurane inhalation will be stopped at the end of surgery.
  Arms: sevoflurane group

SUMMARY:
Postoperative delirium in older adults is a common and costly complication after surgery. Propofol and sevoflurane are commonly used anesthetics to maintain sedation during spine surgery, and have different sedative and anti-inflammatory effects. The aim of this trial will be compare the impact of propofol versus sevoflurane on incidence of postoperative delirium in elderly patients after spine surgery.

DETAILED DESCRIPTION:
Spine surgery is the third most common surgical procedure in older patients. With the increasing number of older patients undergoing spinal surgery, the risk of delirium after spinal surgery is currently expected to increase. The pathophysiological mechanisms of delirium remain poorly understood, leading models include neurotransmitter imbalance and neuroinflammation. Among precipitating factors, drugs (especially sedative hypnotic agents and anticholinergic agents), surgery, anesthesia, high pain levels, anemia, infections, acute illness, and acute exacerbation of chronic illness are the most commonly reported. Propofol and sevoflurane are commonly used anesthetics to maintain sedation during spinal surgery, and induce unconsciousness through different mechanisms. Meanwhile, previous studies have found that propofol and sevoflurane have different anti-inflammatory effects. Given their different sedative and anti-inflammatory effects, propofol and sevoflurane may have different effects on postoperative delirium. There are many studies to explore the effects of propofol and sevoflurane on postoperative delirium, but the conclusions are controversial. Therefore, a randomized, controlled, double-blind clinical study was designed to compare the impact of propofol and sevoflurane on delirium after spine surgery in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥65 years and ≤90 years;
2. scheduled to undergo surgery for spinal, under general anaesthesia;
3. American Society of Anesthesiology (ASA) I-III;
4. agree to participate, and give signed written informed consents.

Exclusion Criteria:

1. family history or history of malignant hyperthermia;
2. History of propofol or sevoflurane allergy;
3. demonstrated cognitive impairment on the modified Mini-Mental State Examination (score, <24of 30 or <20 of 30 if the patient's education year was less than 6 years or<17 if the patient is Illiterate);
4. planned postoperative intubation or transferred to ICU;
5. severe visual or auditory handicap;
6. prior diagnoses of neurologic diseases or mental disorders (e.g., stroke, Parkinson's disease, dementia, schizophrenia, or depressive illness)
7. take anticholinergic drugs or other drugs acting on the central nervous system for a long time before operation
8. participating in other clinical studies in recent 3 months

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium after surgery | Between postoperative day 1 to discharge or day 7, whichever came first
  Delirium is assessed twice daily (8-10 AM and 6-8 PM ) with the 3 minute diagnostic interview for Confusion Assessment Method.Researchers will review all progress notes and nursing documentation for delirium diagnoses, and a thorough medical record review process using the Chart-based Delirium Identification Instrument.

SECONDARY OUTCOMES:
The day of postoperative delirium duration among patients who developed delirium | Time from first to last delirium-positive day. Between postoperative day 1 to discharge or day 7, whichever came first
  Date; Delirium is assessed twice daily (8-10 AM and 6-8 PM ) with the 3 minute diagnostic interview for Confusion Assessment Method
The day of total delirium-positive days among patients who developed delirium | Between postoperative day 1 to discharge or day 7, whichever came first
  Days；Delirium is assessed twice daily (8-10 AM and 6-8 PM ) with the 3 minute diagnostic interview for Confusion Assessment Method
The types of delirium in patients who developed delirium | Between postoperative day 1 to discharge or day 7, whichever came first
  Richmond Agitation- Sedation Scale will be assessed in patients who developed delirium.Patients with delirium are classified into three subtypes: hyperactive (Richmond Agitation Sedation Scale score consistently positive, from +1 to +4), hypoactive (Richmond Agitation Sedation Scale score consistently neutral or negative, from -3 to 0), and mixed.
The intubation time in postanesthesia care unit (PACU) | From the patient transfered into PACU to tracheal extubation. Within 24 hours after surgery.
  minutes
The length of stay in in postanesthesia care unit (PACU) | Within 24 hours after surgery.
  minutes
Incidence of postoperative shivering in PACU | Within 24 hours after surgery.
  Postoperative shivering is assessed in PACU with The Crossley and Mahajan Scale. The Crossley and Mahajan Scale (0 No shivering 1 One or more of the following: piloerection, peripheral vasoconstriction, peripheralcyanosis with no other cause, but no muscle activity 2 Visible muscular activity confined to one muscle group 3 Visible muscular activity in more than one muscle 4 Gross muscular activity involving the whole body).
Postoperative nausea and vomiting | Up to 3 days after surgery
  Postoperative nausea and vomiting is assessed in PACU and postoperative days 1-3(twice daily 8-10 AM and 6-8 PM ).Nausea is defined as a subjective,unpleasant sensation associated with awareness of the urge to vomit. Retching is defined as the laboured, spastic, rhythmic contraction of the respiratory muscles without expulsion of the gastric contents.Vomiting is defined as the forceful expulsion of gastric contents from the mouth. Each episode will be recorded as either present or absent. If the patients had nausea, severity will be recorded using the following scale: 1, mild nausea; 2, moderate nausea; 3, severe nausea. If the patients had retching or vomiting, severity of episodes will be recorded using the following scale: 1, one episode; 2, two episodes; 3, three or more episodes
Incidence of emergence agitation(EA) | Emergence agitation will be assessed immediately after extubation. Within 24 hours after surgery.
  Emergence agitation(EA) is assessed with Richmond Agitation- Sedation Scale (RASS) .The RASS is divided into 10 levels (range of scores, -5 to +4, with higher scores indicating greater agitation). Patients with RASS score > +1 are evaluated as EA
Intensity of pain within 3 days after surgery | Up to 3 days after surgery
  Intensity of pain is assessed twice daily ((8-10 AM and 6-8 PM) with the Visual Analogue Scale ( an 11-point rating scale where 0=no pain and 10=the worst pain )
Postoperative recovery quality | The first day(6-8 PM) after surgery
  Postoperative recovery quality is assessed with Quality of Recovery-40 scale（ QoR40）on the first day(6-8 PM) after surgery.
Length of stay in hospital after surgery | Up to 30 days after surgery
  days
The incidence of non-delirium complications within 30 days after surgery | Up to 30 days after surgery
  The occurrence of non-delirium complications, which are defined as newly occur medical conditions that are harmful for patients' recovery and require therapeutic intervention

CONTACTS AND LOCATIONS:
Overall Officials: wang yuelan, doctor, Study Director — First Affiliated Hospital of Shandong First Medical University,China.
Locations (2):
- China (2):
  - Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University and Shandong Provincial Qianfoshan Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang JH, Lv M, Zhang HX, Gao Y, Chen TT, Wan TT, Wang YL. Impact of propofol versus sevoflurane on the incidence of postoperative delirium in elderly patients after spine surgery: study protocol of a randomized controlled trial. Trials. 2022 Aug 30;23(1):720. doi: 10.1186/s13063-022-06687-x. PMID 36042484